CLINICAL TRIAL: NCT00423163
Title: A Double-Blind, Randomized Controlled Trial of Voriconazole (VFEND®) Plus Micafungin (MYCAMINE™) Versus Voriconazole Plus Placebo in the Treatment of Patients With Proven or Probable Invasive Aspergillosis
Brief Title: A Study to Evaluate the Effectiveness of Voriconazole + Micafungin Versus Voriconazole Alone for Invasive Aspergillosis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: An alternative joint industry effort will provide information on combination versus single agent therapy for treatment of aspergillosis
Sponsor: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-05-002
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Aspergillosis/Blood; Aspergillosis/Invasive
Keywords: Aspergillosis/blood; micafungin; voriconazole; Aspergillus
MeSH Terms: conditions — Aspergillosis | interventions — Micafungin; Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: micafungin
Drug: voriconazole

SUMMARY:
To evaluate the therapeutic effectiveness of voriconazole + micafungin versus voriconazole alone as primary therapy for invasive aspergillosis.

ELIGIBILITY:
Inclusion Criteria:

* Proven, probable or possible invasive aspergillosis
* Patient is 2 years of age or older

Exclusion Criteria:

* The patient has been administered an antifungal agent (voriconazole, itraconazole, posaconazole, caspofungin, micafungin, anidulafungin, amphotericin B, or lipid formulation of amphotericin B) for >7 days immediately prior to randomization for treatment of the Possible, Probable, or Proven invasive aspergillosis for which the patient is being enrolled.
* The patient has been treated with voriconazole for > 7 days immediately prior to randomization

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02

PRIMARY OUTCOMES:
The primary outcome will be Global Success (complete and partial response) at 6 weeks based on the combination of clinical, mycological and radiologic response.

SECONDARY OUTCOMES:
Global Success (GS) at Wk 12, Favorable response (FR) & survival at Wks 6 & 12. GS and FR by infection site, overall frequency of emergent & recurrent fungal infections at Wks 6 & 12, duration of FR, and relationship of galactomannan to clinical outcome

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (44):
- United States (44):
  - Birmingham, Alabama
  - Fountain Valley, California
  - Los Angeles, California
  - Palo Alto, California
  - Sacramento, California
  - San Francisco, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Beech Grove, Indiana
  - Indianapolis, Indiana
  - Kansas City, Kansas
  - Wichita, Kansas
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Boston, Massachusetts
  - Charlestown, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Omaha, Nebraska
  - Albany, New York
  - New York, New York
  - Rochester, New York
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Charlottesville, Virginia
  - Fairfax, Virginia
  - Richmond, Virginia
  - Madison, Wisconsin